CLINICAL TRIAL: NCT02892318
Title: A Phase Ib Study Evaluating the Safety and Pharmacology of Atezolizumab (Anti-PD-L1 Antibody) Administered in Combination With Immunomodulatory Agents in Patients With Acute Myeloid Leukemia
Brief Title: A Study Evaluating the Safety and Pharmacology of Atezolizumab Administered in Combination With Immunomodulatory Agents in Participants With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO30139
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — atezolizumab; guadecitabine

ARMS (4):
- Cohort A1: Safety Cohort (Relapsed/refractory AML) (Experimental): An initial safety evaluation of the combination will be performed in 9 participants with relapsed/refractory AML. All participants will receive atezolizumab (840 milligrams [mg] IV on Days 8 and 22 of every 28-day cycle) administered in combination with guadecitabine (60 milligrams per square meter [mg/m^2] subcutaneously [SC] on Days 1-5 of every 28-day cycle). Treatment with both study drugs will continue until loss of clinical benefit (except in participants who achieve a CR, CRp, or CRi), evidence of unacceptable toxicity, voluntary withdrawal from the study, study termination, or death, whichever occurs first. Participants who achieve a CR, CRp, or CRi will receive an additional six cycles of the combination as consolidation treatment. Participants will discontinue therapy at the end of consolidation response assessment even if the CR, CRp, or CRi is maintained at that time.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine
- Cohort A2: Expansion Cohort (Relapsed/refractory AML) (Experimental): If the combination of atezolizumab and guadecitabine is found to be safe and tolerable in Cohort A1, an expansion cohort of 11 participants with relapsed/refractory AML (Cohort A2) will be evaluated. All participants will receive atezolizumab (840 mg IV on Days 8 and 22 of every 28-day cycle) administered in combination with guadecitabine (60 mg/m^2 SC on Days 1-5 of every 28-day cycle). Treatment with both study drugs will continue until loss of clinical benefit except in participants who achieve a CR, CRp, or CRi), evidence of unacceptable toxicity, voluntary withdrawal from the study, study termination, or death, whichever occurs first. Participants who achieve a CR, CRp, or CRi will receive an additional six cycles of the combination as consolidation treatment. Participants will discontinue therapy at the end of consolidation response assessment even if the CR, CRp, or CRi is maintained at that time.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine
- Cohort A3: Safety Cohort (Previously Untreated AML) (Experimental): If the combination of atezolizumab and guadecitabine is found to be safe and tolerable in Cohort A1, Cohort A3 will assess the safety and tolerability of the combination in 6 participants with untreated AML, who are older and unfit for induction chemotherapy. All participants will receive atezolizumab (840 mg IV on Days 8 and 22 of every 28-day cycle) administered in combination with guadecitabine (60 mg/m^2 SC on Days 1-5 of every 28-day cycle). Treatment with both study drugs will continue until loss of clinical benefit except in participants who achieve a CR, CRp, or CRi), evidence of unacceptable toxicity, voluntary withdrawal from the study, study termination, or death, whichever occurs first. Participants who achieve a CR, CRp, or CRi will receive an additional six cycles of the combination as consolidation treatment. Participants will discontinue therapy at the end of consolidation response assessment even if the CR, CRp, or CRi is maintained at that time.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine
- Cohort A4: Expansion Cohort (Previously Untreated AML) (Experimental): If Cohort A3 is deemed safe and tolerable, an expansion cohort (Cohort A4) of 14 participants with untreated AML, who are older and unfit for induction chemotherapy will be evaluated. All participants will receive atezolizumab (840 mg IV on Days 8 and 22 of every 28-day cycle) administered in combination with guadecitabine (60 mg/m^2 SC on Days 1-5 of every 28-day cycle). Treatment with both study drugs will continue until loss of clinical benefit except in participants who achieve a CR, CRp, or CRi), evidence of unacceptable toxicity, voluntary withdrawal from the study, study termination, or death, whichever occurs first. Participants who achieve a CR, CRp, or CRi will receive an additional six cycles of the combination as consolidation treatment. Participants will discontinue therapy at the end of consolidation response assessment even if the CR, CRp, or CRi is maintained at that time.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 840 mg administered by IV infusion on Days 8 and 22 of each 28-day cycle.
  Other Names: MPDL3280A;; Tecentriq
Drug: Guadecitabine — Guadecitabine 60 mg/m^2 SC on Days 1-5 of every 28-day cycle.

SUMMARY:
This is a non-randomized, open-label, Phase Ib study of atezolizumab in combination with immunomodulatory agents for the treatment of participants with AML (relapsed/refractory and treatment-naive, elderly participants unfit for induction chemotherapy). The study has been designed with the intent, over time, to study multiple combinations of atezolizumab with different immunomodulatory agents in participants with AML. The study will begin with the evaluation of the combination of atezolizumab and guadecitabine (Arm A). In the future, additional arms may be added.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Diagnosis of AML per World Health Organization criteria
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2
* Specifically, for participants in Cohorts A1 and A2: Age greater than or equal to (>=) 18 years, disease progression or failure to achieve complete or partial response after intensive cytotoxic therapy, participants cannot have received more than two prior intensive regimens (e.g., induction + consolidation and one salvage therapy + consolidation)
* Specifically, for participants in Cohorts A3 and A4: Treatment naïve participants unfit for induction chemotherapy for AML as defined by the following: Age >= 70 or age 65 to 69 years with at least one of the following: ECOG performance status of 2, Intermediate I/II or adverse risk cytogenetic and molecular alterations per ELN 2010 guidelines or secondary AML, or other comorbidity judged incompatible with intensive chemotherapy
* Adequate end-organ function
* Willing and able to undergo a pre-treatment bone marrow aspirate and biopsy and subsequent bone marrow aspirates and biopsies during treatment
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 30 days after the last dose of guadecitabine or 5 months after the last dose of atezolizumab, whichever is longer
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* In Cohorts A3 and A4 only, participants with AML eligible for standard intensive induction therapy with an anthracycline and cytarabine
* Prior allogeneic stem cell transplant or solid organ transplant
* Active central nervous system involvement by leukemia
* Pregnant or lactating, or intending to become pregnant during the study
* History of idiopathic pulmonary fibrosis, organizing pneumonitis, drug-induced pneumonitis, idiopathic pneumonitis, or autoimmune disease
* Treatment with investigational therapy within 14 days prior to initiation of study drug
* Any approved AML-related therapy within 14 days prior to enrollment
* Immunosuppressive therapy within 6 weeks of Cycle 1, Day 1
* Daily requirement for corticosteroids (> 10 mg prednisone daily or equivalent) (except for inhalation corticosteroids) within 2 weeks prior to Cycle 1, Day 1
* Prior treatment with immune checkpoint blockade therapies (anti-cytotoxic T-lymphocyte-associated protein 4 [anti-CTLA-4], anti-programmed death-1 [anti-PD-1] or anti-PD-L1) or immune agonists (anti-cluster of differentiation [CD]137, anti-CD40, anti-OX40)
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 half-lives of the drug, whichever is longer, prior to Cycle 1, Day 1
* Treatment with denosumab (or other receptor activator of nuclear factor kappa-B ligand [RANKL] inhibitor) 4 weeks before the first dose and for 10 weeks after the last dose of atezolizumab
* Administration of a live, attenuated vaccine within 4 weeks of Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Planned major surgery during the study
* Positive for hepatitis C virus (HCV) antibody at screening
* Active hepatitis B virus (HBV) infection
* Positive for human immunodeficiency virus (HIV)
* Illicit drug or alcohol abuse within 12 months prior to screening
* Poor peripheral venous access
* Active infection
* Serious infection requiring hospitalization or intravenous (IV) antibiotics within 14 days prior to enrollment
* Any serious medical condition or abnormality in clinical laboratory tests
* History or presence of an abnormal electrocardiogram (ECG)
* History of other malignancy within 2 years prior to screening
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab or guadecitabine formulations
* History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10-31 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to approximately 32 months
Percentage of Participants with Complete Remission (CR) as Defined by International Working Group (IWG) 2003 and European Leukemia Net (ELN) 2010 Response Criteria | After 6 cycles of combination therapy (at Week 24; each cycle is 28 days)
Percentage of Participants with Complete Remission with Incomplete Platelet Recovery (CRp) as Defined by IWG 2003 and ELN 2010 Response Criteria | After 6 cycles of combination therapy (at Week 24; each cycle is 28 days)
Percentage of Participants with Complete Remission with Incomplete Recovery (CRi) as Defined by IWG 2003 and ELN 2010 Response Criteria | After 6 cycles of combination therapy (at Week 24; each cycle is 28 days)
Duration of Response as Defined by IWG 2003 and ELN 2010 Response Criteria | Baseline until the date of relapse/progression or death from any cause, assessed up to approximately 32 months

SECONDARY OUTCOMES:
Percentage of Participants with Best Overall Response as Defined by IWG 2003 and ELN 2010 Response Criteria | Baseline until the date of relapse/progression or death from any cause, assessed up to approximately 32 months
Event-free Survival (EFS) as Defined by IWG 2003 and ELN 2010 Response Criteria | Baseline until the date of induction treatment failure or relapse or death from any cause, assessed up to approximately 32 months
Leukemia-free Survival (LFS) as Defined by IWG 2003 and ELN 2010 Response Criteria | Baseline until the date of relapse or death from any cause, assessed up to approximately 32 months
Overall Survival (OS) | Baseline until death from any cause, assessed up to approximately 32 months
Percentage of Participants with Minimal Residual Disease (MRD) Negativity in Participants who Achieve CR, CRp, or CRi | Baseline up to approximately 32 months
Percentage of Participants with Anti-Drug Antibody (ADA) to Atezolizumab | Pre-infusion (0 hours [hrs]) on Day (D) 1 of Cycle (C) 1; D8 of C2, C3, C4, C6, and every 6 cycles thereafter until treatment discontinuation (up to 32 months); at 120 days and 1 year after atezolizumab last dose (up to 32 months; each cycle is 28 days)
Serum Concentration of Atezolizumab | Day 1 up to 32 months (detailed sample collection time points are provided in Outcome Measure Description)
  Pre-infusion (0 hrs) on D1 of C1, C4; 30 minutes after end of infusion (infusion duration=30-60 minutes) on D8 of C1, C2, C4; Pre infusion (0 hrs) on D22 of C1, D8 of C2, C3, C4, C6, every 6 cycles thereafter until treatment discontinuation (up to 32 months); at 120 days and 1 year after atezolizumab last dose (up to 32 months; each cycle is 28 days)
Plasma Concentration of Guadecitabine | 1, 2, 5, and 8 hours post-injection on D1 of C1 and C4, 1 hour post-injection on D1 of C2, C3, C6, and every 6 cycles thereafter (up to 32 months; each cycle is 28 days)
Plasma Concentration of Decitabine (a Metabolite Product of Guadecitabine) | 1, 2, 5, and 8 hours post-injection on D1 of C1 and C4, 1 hour post-injection on D1 of C2, C3, C6, and every 6 cycles thereafter (up to 32 months; each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Yale University, New Haven, Connecticut
  - The NewYork-Presbyterian Hospital Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - The University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin